CLINICAL TRIAL: NCT00111228
Title: Randomised, Controlled, Multi-centric, Clinical Study to Assess Whether Type 1 Diabetic Patients in Poor Glycemic Control Can Improve Using the Real-time Values of Guardian T Versus Conventional Self-Monitoring Blood Glucose
Brief Title: The Guardcontrol Trial: Study to Assess if Type 1 Diabetics Can Improve Using the Real-time Values of Guardian RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU 007_022004
Record Dates: First submitted 2005-05-18; First posted 2005-05-19 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

ARMS (3):
- Continuous use of the Guardian RT (Experimental): Continuous use of the Guardian RT group
  Interventions: Device: Guardian RT
- Bi-weekly use of the Guardian RT (once every 2 weeks) (Experimental): Bi-weekly use of the Guardian RT (once every 2 weeks) group
  Interventions: Device: Guardian RT
- Control group. SMBG monitoring (Active Comparator): Control group. SMBG monitoring group
  Interventions: Device: SMBG only

INTERVENTIONS:
Device: Guardian RT
  Arms: Bi-weekly use of the Guardian RT (once every 2 weeks); Continuous use of the Guardian RT
Device: SMBG only — SMBG only
  Arms: Control group. SMBG monitoring

SUMMARY:
The objective of the study is to determine whether patients with poor glycemic control can improve metabolic control using the real-time values of the Guardian® RT compared to conventional self-monitoring blood glucose finger-sticks.

DETAILED DESCRIPTION:
Finger-stick based self-testing (SBGM), as well as diagnostic continuous glucose monitoring (CGMS®) allow diabetic patients to find a balance between the two hyper- and hypoglycemic extremes. Nevertheless, there are still patients who fail to achieve good control due to fear of hypoglycemia, or who underestimate post-prandial hyperglycemias.

The Guardian® RT Telemetered Glucose Monitoring System is indicated for continuous or periodic monitoring of real-time interstitial blood glucose values and low/high blood glucose alarms (when pre-set levels are reached) in persons with diabetes mellitus. The glucose values calculated by the device will be used to trigger hypo- and hyperglycemia alerts and will be displayed every 5 minutes. The Guardian® RT stores up to 21 days of data.

The overall primary objective of the study is to determine whether patients with poor glycemic control as evidenced by HbA1c > 8.1% can achieve improved metabolic control using the real-time values of the Guardian® RT compared to conventional self-monitoring blood glucose finger-sticks (control group) after 12 weeks of continuous use.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed Informed consent form prior to Study Entry.
* Patients have been diagnosed with type 1 diabetes mellitus (DM) at least 12 months prior to Study Entry.
* HbA1c must be 8.1% or above at study entry day (central lab value).
* Patients must perform at least two self-monitoring blood glucose finger-sticks daily.
* Patients are on intensive insulin therapy; for multiple daily injections (MDI) patients specifically, be on a schedule of a minimum of 3 injections daily.
* Patients on intensive insulin therapy must be on continuous subcutaneous insulin infusion (CSII) or MDI at least 3 months prior to inclusion and should have been receiving diabetes care from the investigator of each centre for the 6 months prior to inclusion.
* Patients must be using only insulin analogues or rapid-acting human insulin for their meal boluses.
* Patients are willing to undergo all study procedures.
* Patients are trained on how to adapt their insulin dose to their meals and are knowledgeable concerning how to calculate and apply corrective insulin boluses post-prandially, as well as on the influence of physical activity and other life style factors on their glycemia.
* Patients are willing to participate in a Guardian® RT product training course
* Patients understand how to adjust and administer corrective treatment.

Exclusion Criteria:

* Patient has hearing problems/is deaf.
* Patient has impaired vision/blindness so screen alarms cannot be recognized.
* Alcohol or drug abuse other than nicotine.
* Allergy to sensor or components of the sensor.
* Manifest psychiatric disturbances.
* Patients suffering from cancer, heart failure, kidney disease and other chronic debilitating conditions.
* Patient does not have a reliable support person.
* Patient is unwilling or unable to comply with the provisions of the protocol.
* Patient has scheduled travel on a plane in the next 3 months.
* Patient has scheduled a vacation which will occur between Visit 1 and Visit 2.
* Patient is participating in another device or drug study. Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrollment in this trial. The subject may only be enrolled in this study once. Patient has already participated in the Centre Qualification Phase.

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 162 (Actual)
Dates: Start 2004-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee Deiss, MD, Principal Investigator — Klinik für Allgemeine Charité, CVK
Locations (8):
- France (2):
  - Hôpital Sud Francilien, Corbeil Esssonnes
  - CH Robert Debre, Paris
- Klinik für Allgemeine Charité, CVK, Berlin, Germany
- Schneider Children Centre, Petah Tikva, Israel
- Universita Vita-Salute OspedaleS.Raffaele, Milan, Italy
- University Children's Hospital, Ljubljana, Slovenia
- Huddinge University Hospital, Huddinge, Sweden
- Royal Bournemouth Hospital, Bournemouth, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Use of the Guardian RT: Continuous use of the Guardian RT group
  Guardian RT
- Bi-weekly Use of the Guardian RT (Once Every 2 Weeks): Bi-weekly use of the Guardian RT (once every 2 weeks) group
  Guardian RT
Period: Overall Study
Arm/Group | Continuous Use of the Guardian RT | Bi-weekly Use of the Guardian RT (Once Every 2 Weeks) | Control Group. SMBG Monitoring
Started | 54 | 54 | 54
Completed | 49 | 53 | 54
Not Completed | 5 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Use of the Guardian RT | Bi-weekly Use of the Guardian RT (Once Every 2 Weeks) | Control Group. SMBG Monitoring | Total
Number analyzed (Participants) | 54 | 54 | 54 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.24 (13.39) | 25.92 (14.03) | 27.42 (16.53) | 26.52 (14.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 16 | 26 | 71
  Male | 25 | 38 | 28 | 91

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) - Change From Baseline to End of 3 Month Study Period
Description: Hemoglobin A1c (HbA1c) - change from baseline to end of 3 month study period, calculated as A1c at 3 month - A1c at baseline
Time Frame: baseline and 3 month after study
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Arm/Group | Continuous Use of the Guardian RT | Bi-weekly Use of the Guardian RT (Once Every 2 Weeks) | Control Group. SMBG Monitoring
Number analyzed (Participants) | 54 | 54 | 54
percentage of HbA1C | -0.99 (1.13) | -0.70 (1.27) | -0.39 (1.03)

2. Secondary Outcome: Average Blood Glucose - Change From Baseline to End of 3 Month Study Period, Calculated as Average Blood Glucose at 3 Month - Average Blood Glucose at Baseline
Description: Average blood glucose - change from baseline to end of 3 month study period, calculated as average blood glucose at 3 month - average blood glucose at baseline
Time Frame: baseline and 3 month after study
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Continuous Use of the Guardian RT | Bi-weekly Use of the Guardian RT (Once Every 2 Weeks) | Control Group. SMBG Monitoring
Number analyzed (Participants) | 54 | 54 | 54
mg/dL | -12.38 (44.18) | -12.17 (50.37) | -2.21 (45.10)

ADVERSE EVENTS:
Time Frame: 3 month study period
Arm/Group | Continuous Use of the Guardian RT | Bi-weekly Use of the Guardian RT (Once Every 2 Weeks) | Control Group. SMBG Monitoring
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/54 | 2/54 | 2/54
Other Adverse Events (participants affected / at risk) | 15/54 | 15/54 | 10/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Use of the Guardian RT (N=54) | Bi-weekly Use of the Guardian RT (Once Every 2 Weeks) (N=54) | Control Group. SMBG Monitoring (N=54)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatits viral etiology (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ketoacidosis in urinary infection (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
SEVERE HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Acute viral gastroenteritis with DKA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Use of the Guardian RT (N=54) | Bi-weekly Use of the Guardian RT (Once Every 2 Weeks) (N=54) | Control Group. SMBG Monitoring (N=54)
Allergic reaction of the transmitter tape (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bleeding when the 2nd sensor was inserted (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catch a cold and get fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CGMS sensor accidentally pulled out (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fever due to viral syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influence, fever, cough, chest pain (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mild illness with fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mild skin irritation under transmitter tape (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus and redness under the transmitter (General disorders) | 1 (1) | 0 (0) | 0 (0)
Red lesion of toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Redness under the Guardian transmitter (General disorders) | 1 (1) | 0 (0) | 0 (0)
Redness, itching under the sticker for trasmitter (General disorders) | 1 (1) | 0 (0) | 0 (0)
Severe hypo glycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection- viral (Infections and infestations) | 1 (1) | 1 (1) | 5 (6)
Viral gastroenterocolitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Viral upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Minor bleeding at sensor insertion site (General disorders) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Recurrence of upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinopharingitis and fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subperiostal fractute of distal left raduis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Suppurative infection behind right ear (furunculus) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsilopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral rhinopharingitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Otitis with major hyperglycemia for 6 days (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis with major hyperglycemia for 6 days (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach flu (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days